CLINICAL TRIAL: NCT04738487
Title: A Phase 3, Multicenter, Randomized, Double-Blind Study of MK-7684 With Pembrolizumab as a Coformulation (MK-7684A) Versus Pembrolizumab Monotherapy as First Line Treatment for Participants With PD-L1 Positive Metastatic Non-Small Cell Lung Cancer
Brief Title: Coformulation of Pembrolizumab/Vibostolimab (MK-7684A) Versus Pembrolizumab (MK-3475) Monotherapy for Programmed Cell Death 1 Ligand 1 (PD-L1) Positive Metastatic Non-Small Cell Lung Cancer (MK-7684A-003, KEYVIBE-003)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7684A-003; MK-7684A-003 (Other: MSD); jRCT2021210025 (Registry Identifier: jRCT); KEYVIBE-003 (Other: MSD); PHRR230831-006054 (Registry Identifier: PHRR); 2023-505362-28-00 (Registry Identifier: EU CT); U1111-1291-5552 (Registry Identifier: UTN); 2020-004049-35 (EudraCT Number)
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Lung Neoplasms; Non-Small-Cell Lung Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab/Vibostolimab (Experimental): Participants received 200 mg pembrolizumab / 200 mg vibostolimab as a coformulation (MK-7684A) by intravenous (IV) infusion every 3 weeks (Q3W) for up to 35 administrations, until centrally verified disease progression, or until a protocol specified discontinuation criterion was met. Per investigator's discretion, eligible participants with stable disease, or partial/complete response who received a first course treatment may have received a second course of treatment based on original randomization assignment for up to 17 cycles (up to ~1 year).
  Interventions: Biological: Pembrolizumab/Vibostolimab
- Pembrolizumab (Active Comparator): Participants received 200 mg pembrolizumab by IV infusion Q3W for up to 35 administrations, until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met. Per investigator's discretion, eligible participants with stable disease, or partial/complete response who received a first course treatment may have received second course of treatment based on original randomization assignment for up to 17 cycles (up to ~1 year).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab/Vibostolimab — Coformulation of pembrolizumab (MK-3475) 200mg and vibostolimab (MK-7684) 200mg. Participants receive the coformulation by intravenous (IV) infusion every 3 weeks (Q3W) for up to 35 administrations (up to ~2 years).
  Other Names: MK-7684A
  Arms: Pembrolizumab/Vibostolimab
Biological: Pembrolizumab — Participants receive 200 mg of pembrolizumab by intravenous (IV) infusion every 3 weeks (Q3W) for up to 35 administrations (up to ~2 years).
  Other Names: MK-3475; Keytruda
  Arms: Pembrolizumab

SUMMARY:
Researchers are looking for new ways to treat people with metastatic non-small cell lung cancer (NSCLC) that is PD-L1 positive.

* Metastatic means cancer that has spread to other parts of the body.
* PD-L1 positive means that PD-L1 is found on the cancer cells. PD-L1 is a protein that can help the cancer hide from the body's immune system.

The goal of this study is to learn if people who receive vibostolimab and pembrolizumab live longer overall and without the cancer getting worse than people who receive pembrolizumab alone.

DETAILED DESCRIPTION:
The protocol-specified futility analysis of the primary outcome measure was completed with a data cut-off of 05-Sep-2024 (Primary Completion Date) and served as the final analysis of the primary outcome measure. Per protocol, 58 participants enrolled after the primary completion date and will be analyzed in the End of Trial analysis.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of Stage IV: M1a, M1b, or M1c non-small cell lung cancer (NSCLC) per the American Joint Committee on Cancer (AJCC) Staging Manual, version 8
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, as determined by the local site assessment
* Has confirmation that epidermal growth factor receptor (EGFR)-, anaplastic lymphoma kinase (ALK)-, or reactive oxygen species proto-oncogene 1 (ROS1)-directed therapy is not indicated as primary therapy and absence of ALK and ROS1 gene rearrangements
* Has provided tumor tissue that demonstrates Programmed Cell Death 1 Ligand 1 (PD-L1) expression in ≥1% of tumor cells as assessed by immunohistochemistry (IHC) at a central laboratory
* Has an Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1 assessed within 7 days prior to randomization
* Has a life expectancy of at least 3 months
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP)
  * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 120 days after the last dose of study intervention
* Has adequate organ function

Exclusion Criteria:

* Has a known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for at least 3 years since initiation of that therapy
* Has received prior systemic chemotherapy or other targeted or biological antineoplastic therapy for their metastatic NSCLC.

  * Prior treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant or chemoradiation therapy for nonmetastatic NSCLC is allowed as long as therapy was completed at least 6 months before the diagnosis of metastatic NSCLC.
  * Participants must have recovered from all AEs due to previous therapies to Grade ≤1 or baseline. Participants with Grade ≤2 neuropathy may be eligible. Participants with endocrine-related AEs Grade ≤2 requiring treatment or hormone replacement may be eligible.
* Has received prior therapy with an anti-programmed cell death receptor 1 (PD-1), anti-programmed cell death receptor ligand 1 (PD-L1), or anti-programmed cell death receptor ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137)
* Has received previous treatment with another agent targeting the T cell immunoreceptor with immunoglobulin (Ig) and immunoreceptor tyrosine-based inhibition motif (ITIM) domains (TIGIT) receptor pathway
* Has received radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention. Administration of killed vaccines is allowed.

  * Any licensed COVID-19 vaccine (including for Emergency Use) in a particular country is allowed in the study as long as they are mRNA vaccines, adenoviral vaccines, or inactivated vaccines. These vaccines will be treated just as any other concomitant therapy.
  * Investigational vaccines (i.e., those not licensed or approved for Emergency Use) are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has known active or untreated CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable for at least 4 weeks by repeat imaging, clinically stable, and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab/vibostolimab or pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study intervention
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has a known history of interstitial lung disease. Lymphangitic spread of the NSCLC is not exclusionary.
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that prevents the participant from receiving platinum-doublet chemotherapy for first line NSCLC, or that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1264 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2026-01-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (188):
- United States (7):
  - Boca Raton Regional Hospital ( Site 0004), Boca Raton, Florida
  - Illinois Cancer Care ( Site 0026), Peoria, Illinois
  - Mercy Research - Cancer and Hematology Center ( Site 0032), Springfield, Missouri
  - Mercy Research - David C. Pratt Cancer Center ( Site 0025), St Louis, Missouri
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island ( Site 0022), Mineola, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0013), New York, New York
  - Fox Chase Cancer Center-Hematology/Oncology ( Site 0030), Philadelphia, Pennsylvania
- Brazil (8):
  - Hospital São Carlos-Oncocentro Ce ( Site 0208), Fortaleza, Ceará
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0201), Natal, Rio Grande do Norte
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia ( Site 0206), Ijuí, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre-Centro de Pesquisa Novos Tratamentos em Cân, Porto Alegre, Rio Grande do Sul
  - CEPEN - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina ( Site 0209), Florianópolis, Santa Catarina
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA ( Site 0204), Rio de Janeiro
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO-Pesquisa Clinica ( Site 0200), São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo ( Site 0207), São Paulo
- Canada (5):
  - BC Cancer Victoria-Clinical Trials Unit ( Site 0107), Victoria, British Columbia
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0104), Hamilton, Ontario
  - Kingston Health Sciences Centre-Kingston General Hospital Site ( Site 0102), Kingston, Ontario
  - Lakeridge Health ( Site 0106), Oshawa, Ontario
  - Centre Intégré de Santé et de Services Sociaux (CISSS) de La-Centre intégré de cancérologie de Lava, Laval, Quebec
- Chile (11):
  - IC La Serena Research ( Site 0710), La Serena, Coquimbo Region
  - Clínica Puerto Montt ( Site 0713), Port Montt, Los Lagos Region
  - Oncocentro Valdivia ( Site 0715), Valdivia, Los Ríos Region
  - Clinica Universidad Catolica del Maule-Oncology ( Site 0703), Talca, Maule Region
  - Centro de Estudios Clínicos SAGA-CECSAGA ( Site 0712), Santiago, Region M. de Santiago
  - Orlandi Oncologia ( Site 0700), Santiago, Region M. de Santiago
  - FALP ( Site 0702), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0701), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 0711), Temuco, Región de la Araucanía
  - CIDO SpA-Oncology ( Site 0707), Temuco, Región de la Araucanía
  - Bradford Hill Norte ( Site 0708), Antofagasta
- China (30):
  - The First Affiliated Hospital of Anhui Medical University ( Site 2022), Hefei, Anhui
  - Anhui Provincil Hospital South District-Respiratory Medicine Dept ( Site 2017), Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science-Oncology ( Site 2030), Beijing, Beijing Municipality
  - Beijing Cancer hospital-intrathoratic deparmtment II ( Site 2001), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Thoracic Cancer Department A ( Site 2003), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital-pneumology department ( Site 2009), Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University ( Site 2020), Beijing, Beijing Municipality
  - Chongqing Cancer Hospital-Medical Oncology ( Site 2028), Chongqing, Chongqing Municipality
  - Army Medical Center of People's Liberation Army-respiratory ( Site 2025), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital-oncology department ( Site 2023), Fuzhou, Fujian
  - Fuzhou General hospital of Nanjing Military Command-Oncology Department ( Site 2029), Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital-Depatrment of Respiratory and Critical Care Medicine (, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 2006), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 2015), Zhengzhou, Henan
  - Wuhan Union Hospital-Medical Oncology ( Site 2019), Wuhan, Hubei
  - Xiangya Hospital Central South University-Respiratory -Asthma&COPD ( Site 2026), Changsha, Hunan
  - Hunan Cancer Hospital-thoracic oncology II ( Site 2013), Changsha, Hunan
  - Northern Jiangsu People's Hospital-General Surgery Department ( Site 2016), Yangzhou, Jiangsu
  - Jilin Cancer Hospital-oncology department ( Site 2000), Changchun, Jilin
  - Tang Du Hospital ( Site 2004), Xi'an, Shaanxi
  - The First Affiliated Hospital of Xian Jiaotong University wa-Oncology ( Site 2012), Xi'an, Shaanxi
  - LinYi Cancer Hospital ( Site 2034), Linyi, Shandong
  - Linyi People's Hospital-Oncology ( Site 2035), Linyi, Shandong
  - Fudan University Shanghai Cancer Center ( Site 2032), Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University-respiratory ( Site 2018), Chengdu, Sichuan
  - Hangzhou Cancer Hospital-Medical Oncology ( Site 2039), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital-Breast Oncology ( Site 2008), Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University school of medicine-Respiratory Medicine ( Site, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province-Respiratory ( Site 2027), Linhai, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Respiratory department ( Site 2031), Wenzhou, Zhejiang
- Dominican Republic (2):
  - Instituto de Oncologia ( Site 2300), Santo Domingo, Nacional
  - CEMDOE - Centro Médico de Diabetes, Obesidad y Especialidades ( Site 2301), Santo Domingo, Nacional
- Guatemala (6):
  - CELAN,S.A ( Site 0304), Guatemala City
  - Gastrosoluciones ( Site 0302), Guatemala City
  - INTEGRA Cancer Institute ( Site 0303), Guatemala City
  - Onco Go, S.A ( Site 0306), Guatemala City
  - Oncomedica-Guatemala ( Site 0301), Guatemala City
  - Grupo Medico Angeles ( Site 3007), Guatemala City
- Hong Kong (4):
  - Hong Kong Integrated Oncology Centre ( Site 1301), Central
  - Queen Mary Hospital ( Site 1303), Hksar
  - Hong Kong United Oncology Centre ( Site 1302), Jordan
  - Princess Margaret Hospital ( Site 1304), Lai Chi Kok
- Hungary (9):
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház-Megyei Onkológiai Centrum ( Site 1207), Gyula, Bekes County
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 1201), Kecskemét, Bács-Kiskun county
  - Petz Aladar Egyetemi Oktato Korhaz-Pulmonológia ( Site 1205), Győr, Győr-Moson-Sopron
  - Mátrai Gyógyintézet ( Site 1214), Kékestető, Heves County
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Onkologiai Kozpont ( Site 1200), Szolnok, Jász-Nagykun-Szolnok
  - Országos Korányi Pulmonológiai Intézet-XIV. Tüdöbelgyógyászat ( Site 1204), Budapest, Pest County
  - Reformatus Pulmonologiai Centrum-Onkopulmonologiai Jarobeteg Centrum ( Site 1208), Törökbálint, Pest County
  - Zala Megyei Szent Rafael Kórház-Pulmonológia ( Site 1202), Zalaegerszeg, Zala County
  - Semmelweis University-Pulmonológiai Klinika ( Site 1209), Budapest
- India (4):
  - Artemis hospital ( Site 2401), Gurugram, Haryana
  - Tata Memorial Hospital-Medical Oncology ( Site 2404), Mumbai, Maharashtra
  - All India Institute of Medical Sciences ( Site 2403), New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre ( Site 2400), New Delhi, National Capital Territory of Delhi
- Japan (25):
  - National Hospital Organization Nagoya Medical Center ( Site 1920), Nagoya, Aichi-ken
  - Fujita Health University ( Site 1906), Toyoake, Aichi-ken
  - Ehime University Hospital ( Site 1911), Tōon, Ehime
  - Kurume University Hospital ( Site 1912), Kurume, Fukuoka
  - Gunma Prefectural Cancer Center ( Site 1925), Otashi, Gunma
  - National Hospital Organization Hokkaido Cancer Center ( Site 1923), Sapporo, Hokkaido
  - Hyogo College of Medicine-Respiratory Medicine and Hematology ( Site 1922), Nishinomiya, Hyōgo
  - Takarazuka City Hospital ( Site 1924), Takarazuka, Hyōgo
  - Kanagawa Cardiovascular and Respiratory Center ( Site 1921), Yokohama, Kanagawa
  - Kanagawa cancer center ( Site 1916), Yokohama, Kanagawa
  - Sendai Kousei Hospital ( Site 1900), Sendai, Miyagi
  - Niigata Cancer Center Hospital ( Site 1904), Niigata, Niigata
  - Kansai Medical University Hospital ( Site 1914), Hirakata, Osaka
  - Kindai University Hospital- Osakasayama Campus ( Site 1907), Ōsaka-sayama, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center-Department of Thoracic Oncology ( Sit, Sakai, Osaka
  - Osaka Medical and Pharmaceutical University Hospital ( Site 1908), Takatsuki, Osaka
  - Shizuoka Cancer Center ( Site 1905), Nakatogari, Shizuoka
  - Tochigi Cancer Center ( Site 1927), Utsunomiya, Tochigi
  - Chiba University Hospital-Medical Oncology ( Site 1926), Chiba
  - Okayama University Hospital ( Site 1913), Okayama
  - Osaka International Cancer Institute ( Site 1915), Osaka
  - Tokushima University Hospital ( Site 1917), Tokushima
  - Juntendo University Hospital ( Site 1902), Tokyo
  - Japanese Foundation for Cancer Research ( Site 1901), Tokyo
  - Wakayama Medical University Hospital ( Site 1910), Wakayama
- Malaysia (5):
  - University Malaya Medical Centre ( Site 1504), Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan ( Site 1502), Kuantan, Pahang
  - Gleneagles Penang Medical Center-Clinical Research Center (CRC) ( Site 1503), George Town, Pulau Pinang
  - Hospital Pulau Pinang ( Site 1501), George Town, Pulau Pinang
  - National Cancer Institute ( Site 1505), Putrajaya, Putrajaya
- Mexico (9):
  - Actualidad Basada en la Investigación del Cáncer-Lung Cancer ( Site 0411), Guadalajara, Jalisco
  - Arké SMO S.A. de C.V. ( Site 0417), Mexico City, Mexico City
  - Centro de Investigacion Clinica Chapultepec ( Site 0400), Morelia, Michoacán
  - iCan Oncology Center Centro Medico AVE ( Site 0405), Monterrey, Nuevo León
  - Hospital H+ Queretaro ( Site 0416), Querétaro City, Querétaro
  - Medical Care and Research SA de CV ( Site 0409), Mérida, Yucatán
  - Centro Oncologico de Chihuahua-Unidad de Investigacion Clinica ( Site 0402), Chihuahua City
  - Human Science Research Trials ( Site 0406), Mexico City
  - Oaxaca Site Management Organization ( Site 0403), Oaxaca City
- Peru (6):
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 0507), San Isidro, Lima region
  - UNIDAD DE ONCOLOGIA HOSPITAL NACIONAL ADOLFO GUEVARA VELASCO ESSSALUD CUSCO ( Site 0504), Cusco, Qusqu
  - Hospital Guillermo Almenara Irigoyen-Oncology ( Site 0508), Lima
  - Clínica Internacional - Sede San Borja ( Site 0506), Lima
  - INSTITUTO NACIONAL DE ENFERMEDADES NEOPLASICAS ( Site 0500), Lima
  - Hospital Militar Central Luis Arias Schereiber ( Site 0502), Lima
- Philippines (3):
  - East Avenue Medical Center-Department of Medicine ( Site 1605), Quezon City, National Capital Region
  - Veterans Memorial Medical Center-Section of Oncology ( Site 1608), Quezon City, National Capital Region
  - CARDINAL SANTOS MEDICAL CENTER ( Site 1606), San Juan City, Metro Manila, National Capital Region
- Romania (3):
  - Cardiomed SRL Cluj-Napoca ( Site 2201), Cluj-Napoca, Cluj
  - Centrul de Oncologie "Sfântul Nectarie"-Medical Oncology ( Site 2202), Craiova, Dolj
  - SC Medical Center Gral SRL ( Site 2203), Ploieşti, Prahova
- Russia (7):
  - Central Clinical Hospital of the Presidential Administrative Department ( Site 0802), Moscow, Moscow
  - Moscow Regional Oncological Dispensary ( Site 0812), Balashikha, Moscow Oblast
  - Hadassah Medical-Oncology department ( Site 0814), Moscow, Moscow Oblast
  - Nizhegorodsky Regional Oncology Dispensary, Branch #2-chemotherapy ( Site 0809), Nizhny Novgorod, Nizhny Novgorod Oblast
  - GBUZ LOKB-Oncology department #1 ( Site 0804), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary ( Site 0805), Kazan', Tatarstan, Respublika
  - Scientific research institution of oncology named after N.N. Petrov-Thoracic oncology ( Site 0803), Saint Petersburg
- South Africa (8):
  - Wits Clinical Research ( Site 0900), Johannesburg, Gauteng
  - Medical Oncology Centre of Rosebank ( Site 0906), Johannesburg, Gauteng
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 0901), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd-Research ( Site 0902), Sandton, Gauteng
  - Wits Clinical Research-Wits Clinical Research Bara ( Site 0908), Soweto, Gauteng
  - The Oncology Centre ( Site 0905), Durban, KwaZulu-Natal
  - Abraham Oncology ( Site 0907), Richards Bay, KwaZulu-Natal
  - Cape Town Oncology Trials ( Site 0903), Cape Town, Western Cape
- South Korea (10):
  - National Cancer Center-Lung Cancer Center ( Site 1407), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 1403), Seongnam, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Medical Oncology ( Site 1405), Suwon, Kyonggi-do
  - Chungbuk National University Hospital-Internal medicine ( Site 1406), Cheongju-si, North Chungcheong
  - Seoul National University Hospital ( Site 1401), Seoul
  - Kangbuk Samsung Hospital ( Site 1409), Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital-Cancer center ( Site 1410), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 1402), Seoul
  - Asan Medical Center ( Site 1400), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital-Medical Oncology ( Site 1408), Seoul
- Thailand (3):
  - Chulalongkorn University ( Site 1802), Bangkok, Bangkok
  - Ramathibodi Clinical Research Centre ( Site 1801), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 1800), Bangkok, Bangkok
- Turkey (Türkiye) (7):
  - Erciyes University Medical Oncology Department ( Site 1007), Talas, Kayseri
  - Hacettepe Universitesi-oncology hospital ( Site 1001), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 1002), Ankara
  - Gazi Universitesi-Oncology ( Site 1003), Ankara
  - Acıbadem Maslak Hastanesi ( Site 1008), Istanbul
  - Istanbul Universitesi Cerrahpasa-Medical Oncology ( Site 1000), Istanbul
  - Samsun Medical Park Hastanesi-medical oncology ( Site 1005), Samsun
- Ukraine (11):
  - Cherkasy Regional Oncology Dispensary ( Site 1110), Cherkassy, Cherkasy Oblast
  - Chernihiv Medical Center of Modern Oncology-Clinical oncology and gynecology department ( Site 1113), Chernihiv, Chernihiv Oblast
  - Municipal Non-profit Enterprise City Clinical Hospital #4 of Dnipro City Council ( Site 1100), Dnipro, Dnipropetrovsk Oblast
  - MI Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional-Chemotherapy department ( Site 1104), Kryvyi Rih, Dnipropetrovsk Oblast
  - Communal Non-Commercial Enterprise Prykarpatski Clinical Oncological Center of Ivano-Frankivsk Regio, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Institute of General and Emergency Surgery named after V.T. Zaitsev NAMS of Ukraine ( Site 1119), Kharkiv, Kharkivs’ka Oblast’
  - National Cancer Institute ( Site 1114), Kyiv, Kyivska Oblast
  - Vinnytsia Regional Clinical Oncological Hospital ( Site 1102), Vinnytsia, Vinnytsia Oblast
  - Uzhgorod Central City Clinical Hospital-City oncology center ( Site 1120), Uzhhorod, Zakarpattia Oblast
  - Oncolife LLC-day-stay department ( Site 1107), Zaporizhzhia, Zaporizhzhia Oblast
  - Zhytomyr Regional Oncology Center-Chemotherapy Department ( Site 1103), Zhytomyr, Zhytomyr Oblast
- Vietnam (5):
  - Hanoi Oncology Hospital ( Site 2502), Hanoi, Hanoi
  - K Hospital - National Cancer Hospital ( Site 2506), Hanoi, Hanoi
  - National Lung Hospital-Oncology Department ( Site 2503), Hanoi, Hanoi
  - Ho Chi Minh City Oncology Hospital - Tan Phu Ward ( Site 2505), Ho Chi Minh City
  - HCMC University Medical Center-Chemotherapy Department ( Site 2501), Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26159&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Final analysis for the reported results, including participant flow, was performed on 1206 participants enrolled within the primary completion data cutoff. Analysis of the remaining 58 participants will be included in the End of Trial analysis. Per protocol, response/progression or adverse events that occurred during second course were not included in efficacy or safety outcome measures.
Groups:
- Pembrolizumab/Vibostolimab: Participants received 200 mg pembrolizumab / 200 mg vibostolimab as a coformulation (MK-7684A) by intravenous (IV) infusion every 3 weeks (Q3W) for up to 35 administrations, until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met. Per investigator's discretion, eligible participants with stable disease, or partial/complete response who received a first course treatment may have received a second course of treatment based on original randomization assignment for up to 17 cycles (up to ~1 year).
- Pembrolizumab: Participants received 200 mg pembrolizumab by IV infusion Q3W for up to 35 administrations, until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met. Per investigator's discretion, eligible participants with stable disease, or partial/complete response who received a first course treatment may have received a second course of treatment based on original randomization assignment for up to 17 cycles (up to ~1 year).
Period: Overall Study
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab
Started | 594 | 612
Treated | 593 | 610
Received Pembrolizumab/Vibostolimab (MK-7684A) Second Course | 1 | 0
Received Pembrolizumab Second Course | 0 | 3
Completed | 0 | 0
Not Completed | 594 | 612
Not completed — Participant Ongoing in Study | 298 | 297
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 287 | 306

BASELINE CHARACTERISTICS:
Population: Per protocol, analysis population consisted of all participants randomized by the primary completion data cut-off.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab | Total
Number analyzed (Participants) | 594 | 612 | 1206
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (9.8) | 66.3 (10.2) | 66.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 172 | 349
  Male | 417 | 440 | 857
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 152 | 132 | 284
  Not Hispanic or Latino | 434 | 471 | 905
  Unknown or Not Reported | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 28 | 52
  Asian | 247 | 271 | 518
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 291 | 288 | 579
  More than one race | 25 | 22 | 47
  Unknown or Not Reported | 2 | 0 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by ECOG Performance Status. Scores are defined as follows: 0 (Fully active, able to carry on all pre-disease performance without restriction), 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), or 2 (Ambulatory & capable of all selfcare but unable to carry out any work activities, up & about more than 50% of waking hours).
  Participants
    ECOG = 0 | 165 | 163 | 328
    ECOG = 1 | 429 | 448 | 877
    ECOG = 2 | 0 | 1 | 1
Programmed Cell Death Ligand 1 (PD-L1) Status at Baseline [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Randomization of participants in the study was stratified by PD-L1 tumor proportion score (TPS) at baseline (1-49% or ≥ 50%). Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor.
  Participants
    TPS ≥ 50% | 272 | 307 | 579
    TPS 1-49% | 322 | 305 | 627
Geographic Region [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by geographic region of the enrolling site (East Asia vs Non-East Asia).
  Participants
    East Asia | 239 | 260 | 499
    Non-East Asia | 355 | 352 | 707

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants With PD-L1 TPS ≥50%
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to ~39 months
Population: The analysis population consisted of all participants with PD-L1 TPS ≥ 50% who were randomized prior to the primary completion data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab/Vibostolimab: Participants received 200 mg pembrolizumab / 200 mg vibostolimab as a coformulation (MK-7684A) by intravenous (IV) infusion every 3 weeks (Q3W) for up to 35 administrations, until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met.
- Pembrolizumab: Participants received 200 mg pembrolizumab by IV infusion Q3W for up to 35 administrations, until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met.
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab
Number analyzed (Participants) | 272 | 307
Months | 15.7 [12.4 to 24.0] | 20.3 [16.7 to 24.2]
Statistical Analysis 1: Comparison: Pembrolizumab/Vibostolimab vs Pembrolizumab; Test type: Superiority; p = 0.6712, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.83 to 1.35] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

2. Secondary Outcome: OS in Participants With PD-L1 TPS ≥1%
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to ~39 months
Population: The analysis population consisted of all participants with PD-L1 TPS ≥ 1% who were randomized prior to the primary completion data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab
Number analyzed (Participants) | 594 | 612
Months | 15.0 [12.7 to 17.4] | 16.4 [14.9 to 19.1]
Statistical Analysis 1: Comparison: Pembrolizumab/Vibostolimab vs Pembrolizumab; Test type: Superiority; p = 0.3320, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.82 to 1.13] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

3. Secondary Outcome: OS in Participants With PD-L1 TPS 1% to 49%
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Up to ~39 months
Population: The analysis population consisted of all participants with PD-L1 TPS 1% to 49% who were randomized prior to the primary completion data cut-off.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab/Vibostolimab | Pembrolizumab
Number analyzed (Participants) | 322 | 305
Months | 14.3 [11.3 to 17.8] | 14.3 [11.7 to 16.1]
Statistical Analysis 1: Comparison: Pembrolizumab/Vibostolimab vs Pembrolizumab; Test type: Superiority; p = 0.1646, Log Rank — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.72 to 1.11] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

4. Secondary Outcome: Progression-Free Survival (PFS) in Participants With PD-L1 TPS ≥1%
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review will be presented.
Time Frame: Up to ~56 months
Reporting Status: Not Posted

5. Secondary Outcome: PFS in Participants With PD-L1 TPS ≥50%
Description: as for outcome 4
Time Frame: Up to ~56 months
Reporting Status: Not Posted

6. Secondary Outcome: PFS in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 4
Time Frame: Up to ~56 months
Reporting Status: Not Posted

7. Secondary Outcome: Objective Response Rate (ORR) in Participants With PD-L1 TPS ≥1%
Description: ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The percentage of participants who experience a CR or PR as assessed by blinded independent central review based on RECIST 1.1 will be presented.
Time Frame: Up to ~56 months
Reporting Status: Not Posted

8. Secondary Outcome: ORR in Participants With PD-L1 TPS ≥50%
Description: as for outcome 7
Time Frame: Up to ~56 months
Reporting Status: Not Posted

9. Secondary Outcome: ORR in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 7
Time Frame: Up to ~56 months
Reporting Status: Not Posted

10. Secondary Outcome: Duration of Response (DOR) in Participants With PD-L1 TPS ≥50%
Description: For participants who demonstrate a Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by blinded independent central review will be presented.
Time Frame: Up to ~56 months
Reporting Status: Not Posted

11. Secondary Outcome: DOR in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 10
Time Frame: Up to ~56 months
Reporting Status: Not Posted

12. Secondary Outcome: DOR in Participants With PD-L1 TPS ≥1%
Description: as for outcome 10
Time Frame: Up to ~56 months
Reporting Status: Not Posted

13. Secondary Outcome: Change From Baseline in Global Health Status/Quality of Life (QoL) (Items 29, 30) Combined Score on the European Organization for Research and Treatment of Cancer QoL Questionnaire-Core 30 (EORTC QLQ-C30) in Participants With PD-L1 TPS ≥50%
Description: Change from baseline in the score of EORTC QLQ-C30 Items 29 and 30 will be presented. The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

14. Secondary Outcome: Change From Baseline in Global Health Status/QoL (Items 29, 30) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 13
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

15. Secondary Outcome: Change From Baseline in Global Health Status/QoL (Items 29, 30) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 13
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

16. Secondary Outcome: Change From Baseline in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥50%
Description: Change from baseline in the score of EORTC QLQ-C30 Items 1-5 will be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

17. Secondary Outcome: Change From Baseline in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 16
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

18. Secondary Outcome: Change From Baseline in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 16
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

19. Secondary Outcome: Change From Baseline in Role Functioning (Items 6, 7) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥50%
Description: Change from baseline in the score of EORTC QLQ-C30 Items 6-7 will be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

20. Secondary Outcome: Change From Baseline in Role Functioning (Items 6, 7) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 19
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

21. Secondary Outcome: Change From Baseline in Role Functioning (Items 6, 7) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 19
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

22. Secondary Outcome: Change From Baseline in Dyspnea Score (Item 8) on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥50%
Description: Change from baseline in the score of EORTC QLQ-C30 Item 8 will be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

23. Secondary Outcome: Change From Baseline in Dyspnea Score (Item 8) on the EORTC QLQ-C30 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 22
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

24. Secondary Outcome: Change From Baseline in Dyspnea Score (Item 8) on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 22
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

25. Secondary Outcome: Change From Baseline in Cough Score (Item 31) on the European Organization for Research and Treatment of Cancer Quality of Life Lung Cancer-Specific Questionnaire Module (EORTC QLQ-LC13) in Participants With PD-L1 TPS ≥50%
Description: Change from baseline in the score of EORTC QLQ-LC13 Item 31 will be presented. The EORTC QLQ-LC13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates more frequent coughing
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

26. Secondary Outcome: Change From Baseline in Cough Score (Item 31) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 25
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

27. Secondary Outcome: Change From Baseline in Cough Score (Item 31) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 25
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

28. Secondary Outcome: Change From Baseline in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS ≥50%
Description: Change from baseline in the score of EORTC QLQ-LC13 Item 40 will be presented. The EORTC QLQ-LC13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of chest pain.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

29. Secondary Outcome: Change From Baseline in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 28
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

30. Secondary Outcome: Change From Baseline in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 28
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

31. Secondary Outcome: Time to Deterioration (TTD) in Global Health Status/QoL (Items 29, 30) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥50%
Description: TTD in the score of EORTC QLQ-C30 Items 29 and 30 will be presented. The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

32. Secondary Outcome: TTD in Global Health Status/QoL (Items 29, 30) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 31
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

33. Secondary Outcome: TTD in Global Health Status/QoL (Items 29, 30) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 31
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

34. Secondary Outcome: TTD in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥50%
Description: TTD in the score of EORTC QLQ-C30 Items 1-5 will be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

35. Secondary Outcome: TTD in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1% to 49%
Description: as for outcome 34
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

36. Secondary Outcome: TTD in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 34
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

37. Secondary Outcome: TTD in Role Functioning (Items 6, 7) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥50%
Description: TTD in the score of EORTC QLQ-C30 Items 6-7 will be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

38. Secondary Outcome: TTD in Role Functioning (Items 6, 7) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 37
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

39. Secondary Outcome: TTD in Role Functioning (Items 6, 7) Combined Score on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 37
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

40. Secondary Outcome: TTD in Dyspnea Score (Item 8) on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥50%
Description: TTD in the score of EORTC QLQ-C30 Item 8 will be presented. The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

41. Secondary Outcome: TTD in Dyspnea Score (Item 8) on the EORTC QLQ-C30 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 40
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

42. Secondary Outcome: TTD in Dyspnea Score (Item 8) on the EORTC QLQ-C30 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 40
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

43. Secondary Outcome: TTD in Cough Score (Item 31) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS ≥50%
Description: TTD in the score of EORTC QLQ-LC13 Item 31 will be presented. The EORTC QLQ-LC13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates more frequent coughing. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

44. Secondary Outcome: TTD in Cough Score (Item 31) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 43
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

45. Secondary Outcome: TTD in Cough Score (Item 31) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 43
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

46. Secondary Outcome: TTD in in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS ≥50%
Description: TTD in the score of EORTC QLQ-LC13 Item 40 will be presented. The EORTC QLQ-LC13 is a lung cancer specific health-related quality-of life (QoL) questionnaire. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of chest pain. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

47. Secondary Outcome: TTD in in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS 1% to 49%
Description: as for outcome 46
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

48. Secondary Outcome: TTD in in Chest Pain Score (Item 40) on the EORTC QLQ-LC13 in Participants With PD-L1 TPS ≥1%
Description: as for outcome 46
Time Frame: Baseline and up to ~56 months
Reporting Status: Not Posted

49. Secondary Outcome: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: The number of participants who experienced an adverse event (AE) will be presented. An AE is defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to ~56 months
Reporting Status: Not Posted

50. Secondary Outcome: Number of Participants Who Discontinued Study Intervention Due to an Adverse Event (AE)
Description: The number of participants who discontinue study intervention due to an adverse event (AE) will be presented. An AE is defined as any untoward medical occurrence in a participant administered study treatment and which did not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to ~56 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 39 months
Description: Serious & Other AEs include participants randomized by primary completion data cutoff who received ≥1 dose of study drug. All-Cause Mortality (ACM) includes participants randomized by primary completion data cutoff. Progression of cancer was not deemed an AE unless related to study treatment. MedDRA terms "Neoplasm progression" "Malignant neoplasm progression" & "Disease progression" not related to study treatment are excluded as AEs. ACM & AEs reported separately for second course treatment.
Groups:
- Pembrolizumab/Vibostolimab First Course: Participants received 200 mg pembrolizumab / 200 mg vibostolimab as a coformulation (MK-7684A) by intravenous (IV) infusion every 3 weeks (Q3W) for up to 35 administrations, until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met.
- Pembrolizumab First Course: Participants received 200 mg pembrolizumab by IV infusion Q3W for up to 35 administrations, until centrally verified disease progression, or until a protocol-specified discontinuation criterion was met.
- Pembrolizumab/Vibostolimab Second Course: Participants who stopped pembrolizumab/vibostolimab after receiving 35 treatment cycles or participants who stopped pembrolizumab/vibostolimab after attaining a confirmed CR were eligible for a second course of pembrolizumab/vibostolimab. Participants received 200 mg pembrolizumab / 200 mg vibostolimab as a coformulation (MK-7684A) by IV infusion Q3W for up to 17 additional administrations.
- Pembrolizumab Second Course: Participants who stopped pembrolizumab after receiving 35 treatment cycles or participants who stopped pembrolizumab after attaining a confirmed CR were eligible for a second course of pembrolizumab. Participants received 200 mg pembrolizumab by IV infusion Q3W for up to 17 additional administrations.
Arm/Group | Pembrolizumab/Vibostolimab First Course | Pembrolizumab First Course | Pembrolizumab/Vibostolimab Second Course | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 291/594 | 310/612 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 249/593 | 220/610 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 478/593 | 472/610 | 1/1 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab/Vibostolimab First Course (N=593) | Pembrolizumab First Course (N=610) | Pembrolizumab/Vibostolimab Second Course (N=1) | Pembrolizumab Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Myocardial injury (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 10 (10) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 6 (6) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mycoplasma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 57 (66) | 56 (60) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 7 (7) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (12) | 8 (8) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bone callus excessive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral microinfarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 5 (6) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myelitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Immune-mediated cystitis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchus compression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (7) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 12 (14) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 8 (8) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SJS-TEN overlap (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical aid in dying (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab/Vibostolimab First Course (N=593) | Pembrolizumab First Course (N=610) | Pembrolizumab/Vibostolimab Second Course (N=1) | Pembrolizumab Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 145 (182) | 117 (162) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 39 (50) | 29 (32) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 56 (74) | 67 (78) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 65 (76) | 59 (66) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 51 (68) | 59 (84) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 67 (81) | 45 (48) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 30 (33) | 20 (24) | 0 (0) | 0 (0)
Fatigue (General disorders) | 61 (70) | 62 (69) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 59 (69) | 38 (40) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 52 (58) | 51 (54) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 34 (37) | 35 (36) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 17 (18) | 39 (51) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 32 (36) | 27 (35) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 73 (98) | 72 (100) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 46 (76) | 43 (56) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 78 (96) | 79 (106) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 43 (58) | 32 (35) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 28 (41) | 45 (54) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 31 (49) | 23 (29) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 39 (59) | 37 (46) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 72 (80) | 69 (77) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 21 (31) | 9 (17) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 74 (82) | 84 (93) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 44 (70) | 44 (67) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 69 (89) | 73 (98) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 32 (45) | 28 (44) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 52 (74) | 52 (67) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 (53) | 49 (58) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 35 (37) | 38 (41) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 51 (54) | 69 (73) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 (47) | 53 (57) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 32 (35) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 38 (45) | 14 (15) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 106 (128) | 57 (69) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 92 (116) | 53 (78) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 31 (36) | 20 (31) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04738487/Prot_SAP_000.pdf